CLINICAL TRIAL: NCT04879771
Title: Comparison of Receiving Painless Gastrointestinal Endoscopy in the Morning or Afternoon on Postoperative Sleep Quality
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Yanchao Yang, principal investigator, Shengjing Hospital
Other Study IDs: GIE and sleep
Record Dates: First submitted 2021-05-07; First posted 2021-05-10 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Morning Inspections; Afternoon Inspections; Sleep Quality; Gastrointestinal Endoscopy; Pain; General Anesthesia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Morning GIE
  Interventions: Procedure: Receive gastrointestinal endoscopy
- Afternoon GIE
  Interventions: Procedure: Receive gastrointestinal endoscopy

INTERVENTIONS:
Procedure: Receive gastrointestinal endoscopy — patients receive gastrointestinal endoscopy in the morning or afternoon

SUMMARY:
Gastrointestinal endoscopy (GIE) are important examinations for screening, diagnosing, and treating a variety of gastrointestinal diseases. Specifically, endoscopy is one of the best surveillance tools for early detection of several cancers, GIE is increasingly being used because of government support for cancer screening and growing interest in preventive medicine. But some patients refuse endoscopic examinations because of fear and anxiety of discomfort during the procedure. Sedatives is increasingly used in GIE these years to reduce the anxiety and discomfort of patients and increase patient satisfaction. Sedatives also minimize the risk of patient injury during GIE and provide ideal working conditions for endoscopists to improve patients' satisfaction with surgery. Sedation can be divided into four levels: minimal sedation (anxiolysis), conscious sedation, deep sedation, and general anesthesia. A combination of benzodiazepines and opiates (midazolam and fentanyl), the medications used most commonly by gastroenterologists for procedural sedation, provides adequate analgesia and sedation during colonoscopy. Besides above, propofol is an intravenously administered hypnotic drug used for induction and maintenance of general anaesthesia and is also used in procedural sedation. Nowadays, propofol sedation is preferred by more and more endoscopists for colonoscopy procedures with its perceived benefits of rapid postprocedure drug clearance, improved patient comfort and rapid recovery/discharge when compared to conventional sedation. And propofol provided more rapid recovery than midazolam, it has the merit of post-procedure neuropsychologic function over midazolam. Previous studies have found that general anesthesia, as an independent risk factor, may lead to desynchronization of the circadian rhythm, which could result in postoperative sleep disorders characterized by reduced rapid eye movement (REM) and slow-wave sleep (SWS). Postoperative sleep disorders could cause serious adverse effects on postoperative outcomes, such as postoperative fatigue, severe anxiety and depression, emotional detachment and delirium, and even increased pain sensitivity or postoperative pain in patients. Previous studies have found that general anesthesia, as an independent risk factor, may lead to desynchronization of the circadian rhythm, which could result in postoperative sleep disorders characterized by reduced rapid eye movement (REM) and slow-wave sleep (SWS). Postoperative sleep disorders could cause serious adverse effects on postoperative outcomes, such as postoperative fatigue, severe anxiety and depression, emotional detachment and delirium, and even increased pain sensitivity or postoperative pain in patients. At present, there are few studies that have assessed the effect of circadian rhythm during different timings of gastrointestinal endoscopy on postoperative sleep quality, and pain under general anesthesia.

Based on these considerations, we sought to answer the questions in this study:

1. What is the impact of morning operation and evening operation on the intraoperative anesthetic requirement under general anesthesia?
2. What are the effects of different timings of surgery on the postoperative sleep quality and pain under general anesthesia?

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 65 years,
* ASA physical status of I or II.

Exclusion Criteria:

* presence of sleep disorders
* pain syndrome
* cardiovascular disease
* sleep apnea syndrome
* psychosis
* history of opioid usage
* history of abnormal operation or anesthesia recovery
* unwillingness to provide informed consent
* patient with a language communication disorder.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received gastrointestinal endoscopy under general anesthesia at Shengjing Hospital of China Medical University were enrolled in this study
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-05-07 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
postoperative sleep quality | first night after inspections
  assess sleep quality by using the Athens insomnia scale Total AIS scores range from 0 to 24 points. A total score of ≥ 6 points indicates a diagnosis of insomnia
postoperative sleep quality | second night after inspections
  assess sleep quality by using the Athens insomnia scale Total AIS scores range from 0 to 24 points. A total score of ≥ 6 points indicates a diagnosis of insomnia

SECONDARY OUTCOMES:
postoperative pain score | 24 hours after surgery
  assess pain level by using VAS score Postoperative pain scores were evaluated by the visual analog scale (VAS) score,15 where 0 indicates painlessness, and 10 indicates severe pain. The VAS score was measured at 1, 6, 12, and 24 hours postoperatively
postoperative adverse effects | 24 hours after surgery
  assess postoperative adverse effects

CONTACTS AND LOCATIONS:
Overall Officials: Junchao Zhu, Study Director — Shengjing Hospital
Locations (1):
- Shengjing Hospital, Shenyang, Liaoning, China